CLINICAL TRIAL: NCT06847399
Title: Efficacy and Safety of Tirzepatide Versus Placebo or Lisdexamfetamine Dimesylate for Binge-Eating Disorder: A Randomized Clinical Trial
Brief Title: Efficacy and Safety of Tirzepatide Versus Placebo or Lisdexamfetamine Dimesylate for Binge-Eating Disorder
Acronym: LIBERATE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00474917
Record Dates: First submitted 2025-02-24; First posted 2025-02-26 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Obesity and Overweight; Binge Eating Disorder
Keywords: obesity; binge eating disorder; tirzepatide; Lisdexamfetamine
MeSH Terms: conditions — Obesity; Overweight; Binge-Eating Disorder | interventions — Tirzepatide; Lisdexamfetamine Dimesylate; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Tirzepatide (Experimental): Tirzepatide injection + placebo oral capsule
  Interventions: Drug: Tirzepatide; Behavioral: Guided self-help cognitive behavioral therapy; Drug: Placebo (oral)
- Lisdexamfetamine dimesylate (Active Comparator): Placebo injection + lisdexamfetamine dimesylate
  Interventions: Drug: Lisdexamfetamine Dimesylate; Behavioral: Guided self-help cognitive behavioral therapy; Drug: Placebo (injection)
- Placebo (Placebo Comparator): Placebo injection + placebo oral capsule
  Interventions: Behavioral: Guided self-help cognitive behavioral therapy; Drug: Placebo (oral); Drug: Placebo (injection)

INTERVENTIONS:
Drug: Tirzepatide — Tirzepatide
  Arms: Tirzepatide
Drug: Lisdexamfetamine Dimesylate — Lisdexamfetamine dimesylate
  Arms: Lisdexamfetamine dimesylate
Behavioral: Guided self-help cognitive behavioral therapy — Guided self-help cognitive behavioral therapy
Drug: Placebo (oral) — Placebo (oral)
  Arms: Placebo; Tirzepatide
Drug: Placebo (injection) — Placebo (injection)
  Arms: Lisdexamfetamine dimesylate; Placebo

SUMMARY:
The purpose of this study is to assess the efficacy and safety of tirzepatide in adults with obesity and binge-eating disorder, comparing tirzepatide against placebo and lisdexamfetamine dimesylate. All participants will receive guided self-help cognitive behavioral therapy.

ELIGIBILITY:
Inclusion Criteria:

Disease Characteristics

1. Have a BMI ≥30 kg/m2 or ≥27 kg/m2

   * previously diagnosed with at least one obesity-related comorbidity:
2. Have at least one self-reported unsuccessful dietary effort to lose body weight
3. Meet Diagnostic and Statistical Manual (DSM)-5 criteria for Binge Eating Disorder (BED) as diagnosed by the Eating Disorder Examination interview and confirmed by binge-eating diaries that is moderate or greater in severity (4 or more episodes per week)

   Participant Characteristics
4. Are 18 years of age or older
5. Participants assigned female at birth: (participants assigned female at birth who are not of childbearing potential may participate and include those who are:

   * infertile due to surgical sterilization (hysterectomy, bilateral oophorectomy or tubal ligation), congenital anomaly such as Mullerian agenesis
   * postmenopausal, defined as either
   * a female at least 40 years of age with an intact uterus, not on hormone therapy and who has cessation of menses for at least 1 year without an alternative medical cause; women in this category must test negative in pregnancy test prior to study entry OR
   * a female 55 or older not on hormone therapy, who has had at least 12 months of spontaneous amenorrhea OR
   * a female at least 55 years of age with a diagnosis of menopause prior to starting hormone replacement therapy

   Participants assigned female at birth of child-bearing potential (not surgically sterilized and between menarche and 1-year postmenopausal) must:
   * test negative for pregnancy at Visit 1 based on a serum pregnancy test
   * and if sexually active, agree in writing to use 2 forms of effective contraception, where at least 1 form is highly effective, for the duration of the trial
   * not be breastfeeding

   Informed Consent
6. Understand and be willing to comply with all study-related procedures and agree to participate in the study by giving written informed consent in accordance with local regulations
7. In the investigator's opinion, are well-motivated, capable, and willing to:

   * Learn how to self-inject study drug, as required for this protocol (persons with visual impairments or physical limitations who are not able to perform the injections must have the assistance of an individual trained to inject study drug)
   * Inject study drug (or receive an injection from a trained individual if visually impaired or with physical limitations)
   * Learn how to take oral capsules, be consistently able to swallow capsules, and willing to take oral capsules daily as required for this protocol
   * Follow study procedures for the duration of the study

   Exclusion Criteria:

   Medical Conditions

   Eating disorder-related
8. Current diagnosis of bulimia nervosa or anorexia nervosa

   Diabetes-related
9. Have type 1 diabetes mellitus (T1DM) or Type 2 diabetes mellitus (T2DM), history of ketoacidosis, or hyperosmolar state/coma
10. Have laboratory evidence diagnostic of diabetes mellitus during screening, including an HbA1c ≥6.5% or fasting glucose >126 mg/dL

    Obesity-related:
11. Have a self-reported change in body weight >5 kg within 3 months prior to screening
12. Have a prior or planned surgical treatment for obesity (excluding lap-band if removed >6 months prior to screening or liposuction or abdominoplasty if performed >1 year prior to screening)
13. Have or plan to have endoscopic and/or device-based therapy for obesity or have had device removal within the last 6 months prior to screening (for example, mucosal ablation, gastric artery embolization, intragastric balloon and duodenal-jejunal bypass sleeve)

Other medical

* Have a family or personal history of medullary thyroid carcinoma (MTC) or Multiple Endocrine Neoplasia (MEN) Syndrome type 2
* Known serious hypersensitivity to tirzepatide or lisdexamfetamine dimesylate or any of the excipients in the medications
* Have severe gastrointestinal disease
* Have known clinically significant renal impairment
* Have uncontrolled medical conditions or contraindications to tirzepatide or lisdexamfetamine dimesylate
* Have personal or family history of cardiovascular disease that could increase vulnerability to sympathomimetic effects of psychostimulants
* Have a history of suspected substance abuse within the past 5 years
* Have a lifetime history of psychostimulant abuse and/or dependence
* Have glaucoma
* Have had a history of chronic or acute pancreatitis
* Have obesity induced by other endocrinologic disorders (for example, Cushing Syndrome) or diagnosed monogenetic or syndromic forms of obesity (for example, Melanocortin 4 Receptor deficiency or Prader Willi Syndrome)
* Have a current diagnosis of attention-deficit/hyperactivity disorder
* Have a history of significant active or unstable Major Depressive Disorder (MDD; within the last 2 years) or other severe psychiatric disorder (for example, schizophrenia, bipolar disorder, psychosis, mania, hypomania, or other serious mood or anxiety disorder) Note: Patients with MDD or generalized anxiety disorder whose disease state is considered stable and expected to remain stable throughout the course of the study, in the opinion of the investigator, may be considered for inclusion if not on excluded medications
* Have a Patient Health Questionnaire-9 (PHQ-9) score of 15 or more at Visit 1 or 2, prior to randomization
* Have any lifetime history of a suicide attempt
* Individual is considered a suicide risk in the opinion of the investigator; or endorsement of current, active suicidal ideation at screening or randomization. On the Columbia-Suicide Severity Rating Scale (C-SSRS) at Visits 1 or 2, prior to randomization:

  * a "yes" answer to either Question 4 (Active Suicidal Ideation with Some Intent to Act, Without Specific Plan) or
  * a "yes" answer to Question 5 (Active Suicidal Ideation with Specific Plan and Intent) on the "Suicidal Ideation" portion of the C-SSRS or
  * a "yes" answer to any of the suicide-related behaviors (Actual Attempt, Interrupted Attempt, Aborted Attempt, Preparatory Act or Behavior) on the "Suicidal Behavior" portion of the C-SSRS and
  * the ideation or behavior occurred within the past month
* Have taken monoamine oxidate inhibitors (MAOI), or within 14 days of stopping MAOIs
* Have uncontrolled hypertension (SBP above or equal to 160 mmHg and/or diastolic blood pressure above or equal to 100 mmHg)
* Have any of the following cardiovascular conditions within 3 months prior to randomization: acute myocardial infarction (MI), cerebrovascular accident (stroke), unstable angina
* Have a history of an active or untreated malignancy or are in remission from a clinically significant malignancy (other than basal- or squamous-cell skin cancer, in situ carcinomas of the cervix, or in situ prostate cancer) for less than 5 years
* History of seizures (other than infantile febrile seizures), any tic disorder, or a current diagnosis and/or known family history of Tourette's Disorder, serious neurological disease, history of significant head trauma, dementia, Parkinson's disease, or intracranial lesions
* Participant has known history of symptomatic cardiovascular disease, advanced arteriosclerosis, structural cardiac abnormality, cardiomyopathy, serious heart rhythm abnormalities, coronary artery disease, or other serious cardiac problems that may place the participant at increased vulnerability to the sympathomimetic effects of a stimulant medication
* Have a history of any other condition that, in the opinion of the investigator, may preclude the participant from following and completing the protocol

Prior/Concomitant Therapy

* Are receiving concurrent treatment for eating or weight disorders
* Use of a psychostimulant within the past 6 months
* Have taken within 3 months prior to screening, medications (prescribed or over-the counter) intended to promote weight loss. Examples include, but are not limited to

  * Saxenda® (liraglutide 3.0 mg)
  * Xenical®/Alli® (orlistat)
  * Meridia® (sibutramine)
  * Adipex® (phentermine)
  * BELVIQ® (lorcaserin)
  * Qsymia® (phentermine/topiramate combination)
  * Contrave® (naltrexone/bupropion)
  * Ozempic or Wegovy (semaglutide)
  * Mounjaro or Zepbound (tirzepatide)
  * Rybelsus (semaglutide)

Prior/Concurrent Clinical Study Experience

* Are currently enrolled in any other clinical study involving an investigational product (IP) or any other type of medical research judged not to be scientifically or medically compatible with this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2025-09-17 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Percent initial weight loss | Baseline to 52 weeks
  To compare tirzepatide maximum tolerated dose (MTD) versus placebo from randomization to week 52 for percent initial weight loss
Change in the Number of Binge-eating episodes | Baseline to 52 weeks
  To compare tirzepatide MTD versus placebo from randomization to week 52 for reduction in the number of binge-eating episodes defined as change in the number of binge-eating episodes in the past 28 days measured via clinician interview

SECONDARY OUTCOMES:
Number of Binge-eating episodes | Baseline to 52 weeks
  To assess the non-inferiority of tirzepatide MTD versus lisdexamfetamine dimesylate MTD from randomization to week 52 for reduction in the number of binge-eating episodes defined as change in the number of binge-eating episodes in the past 28 days measured via clinician interview
Percentage of Participants Achieving Binge-eating abstinence | Baseline to 52 weeks
  To compare tirzepatide MTD versus placebo from randomization to week 52 for binge-eating abstinence, defined as percent of study participants who achieve 0 episodes of binge eating in the past 28 days via clinician interview
Number of Participants who achieve ≥5% body weight reduction | Baseline to 52 weeks
  To compare tirzepatide MTD versus placebo from randomization to week 52 for percent of study participants who achieve ≥5% body weight reduction. Categorical achievement of weight reduction threshold (≥5% initial weight loss).
Number of Participants who achieve ≥10% body weight reduction | Baseline to 52 weeks
  To compare tirzepatide MTD versus placebo from randomization to week 52 for percent of study participants who achieve ≥10% body weight reduction. Categorical achievement of weight reduction threshold (≥10% initial weight loss)
Number of Participants who achieve ≥15% body weight reduction | Baseline to 52 weeks
  To compare tirzepatide MTD versus placebo from randomization to week 52 for percent of study participants who achieve ≥15% body weight reduction. Categorical achievement of weight reduction threshold (≥15% initial weight loss)
Number of Participants who achieve ≥20% body weight reduction | Baseline to 52 weeks
  To compare tirzepatide MTD versus placebo from randomization to week 52 for percent of study participants who achieve ≥20% body weight reduction. Categorical achievement of weight reduction threshold (≥20% initial weight loss).
Clinical global functioning as assessed by the Clinical Global Impressions Scale (CGI) score | Baseline to 52 weeks
  To compare tirzepatide MTD versus placebo from randomization to week 52 for clinical global functioning using change in Clinical Global Impressions Scale (CGI) score. The CGI severity scale rates the severity of a participant's condition (range: 1 [normal, not at all ill] to 7 [among the most extremely ill]). The CGI improvement scale rates overall symptom improvement in the participant's condition relative to baseline (range: 1 [very much improved] to 7 [very much worse]). Score range 0-21. Higher score worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ariana M Chao, PhD, CRNP, FNP-BC, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States